CLINICAL TRIAL: NCT05534542
Title: Comparison of the Effectiveness of Intradialytic Core Stabilization and Aerobic Exercise in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: cngztaskaya
Record Dates: First submitted 2022-09-01; First posted 2022-09-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-03

CONDITIONS: Hemodialysis Complication
Keywords: hemodialysis; dialysis efficiency; fatigue; quality of life; sleep; functionality
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stabılızatıon (Active Comparator): use of ıntradıalıtıc core stabılızatıon ın hemodıalysıs patıents
  Interventions: Other: exercıse
- aerobıc exercıse (Active Comparator): use of ıntradıalıtıc aerobıc exercıse ın hemodıalysıs patıents
  Interventions: Other: exercıse

INTERVENTIONS:
Other: exercıse — ıntradıalıtıc core stabılızatıon

SUMMARY:
Purpose: To examine the effects of core stabilization and aerobic exercises on dialysis adequacy, functionality level, and quality of life in hemodialysis (HD) patients. The secondary aim of the study is to compare the effectiveness of intradialytic core stabilization and aerobic exercises in HD patients.

Materials and Methods: Patients who received hemodialysis treatment for 4 hours, 3 days a week were planned to be included in this randomized controlled study. Patients participating in the study will be randomly divided into 2 groups. Grup 1 was planned to be given core stabilization exercises during hemodialysis three times a week for eight weeks; Group 2 was planned to be given aerobic exercise during hemodialysis three times a week for eight weeks. It aimed to evaluate the patients in the weeks before the start of the treatment and the week after the end of the treatment. Personal information form for evaluation, dialysis adequacy, quality of life questionnaire-kidney disease quality of life-36, piper fatigue scale, hospital anxiety and depression scale (hads), Pittsburgh sleep scale, five times sit and stand test, 10 m walking test , tinetti balance and walking test, and 2-minute step test were planned to be used.

ELIGIBILITY:
Inclusion Criteria:

* To receive HD treatment for a minimum of 6 months, for 4 hours per day, three days per week
* Being 18 years or older
* A score of 3 and/or below in the Sarcopenia Screening Test (SARC-F)

Exclusion Criteria:

* Having a history of myocardial infarction in the last 3 months
* Having angina pectoris, arrhythmia, or uncontrolled hypertension
* Having communication and/or cognitive issues that prevent them from meeting the requirements of the tests
* Becoming pregnant or going through infertility treatment
* Having a psychiatric diagnosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Dialysis adequacy | one month
  Dialysis adequacy is determined as the urea reduction rate (URR) and unitless Kt/V value. In calculating the Kt/V value; K-is the urea clearance coefficient of the dialyzer (ml/min), t refers to dialysis time (min), and V signifies the urea distribution volume (ml).
Kidney Disease Quality of Life-36 (KDQOL-36) | Two months
  The KDQOL-36 is a measure of kidney disease-related quality of life that comprises four subscales: generic core [Physical Component Summary (PCS, 12 items) and Mental Component Summary (MCS, 12 items)]; Symptoms/Problems (12 items); Burden of Kidney Disease (4 items), and Effects of Kidney Disease (8 items).
Five times sit-to-stand test | Two months
  The Five-Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements.
2 Minute Step Test | Two months
  The test, known as the 2-minute step test (TMST), simply requires that tested individuals march in place as fast as possible for 2 minutes while lifting their knees to a height midway between their patella and iliac crest when standing.
10 Metre Walk Test | Two months
  The 10 meter walk test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.

SECONDARY OUTCOMES:
Piper Fatigue Scale | Two months
  The Piper Fatigue Scale (PFS) is one of the commonly used multidimensional fatigue measures and includes subdomains of behavioral, affective, sensory, and cognitive/mood attributes of fatigue.
Hospital Anxiety and Depression Scale (HADS) | Two months
  The HADS was developed to detect states of anxiety and depression in hospitalized patients. The measure was designed to exclude items that might conflate anxiety or depression with physical health problems.
Pittsburgh Sleep Quality Index (PSQI) | Two months
  PSQI is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval.
Tinetti Gait and Balance Test | Two months
  The Tinetti assessment tool is an easily administered, task-oriented test that measures an adult's gait and balance abilities. To assess balance, the patient is seated in a firm, armless chair. stand next to the patient to evaluate the gait. The patient is asked to walk normally and then speed up.

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz TAŞKAYA, Principal Investigator — scholar; Buket Büyükturan, Study Director — scholar
Locations (1):
- Mus State Hospital, Muş, Muş, Turkey (Türkiye)